CLINICAL TRIAL: NCT03969693
Title: A Prospective Observational Study With Longitudinal Cardiopulmonary Surveillance in Lymphoma Patients Undergoing Mediastinal Radiotherapy in the Era of Modern Chemoradiation
Brief Title: Lymphoma Patients Undergoing Mediastinal Radiotherapy in the Era of Modern Chemoradiation
Status: Not yet recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1810020038
Record Dates: First submitted 2019-05-26; First posted 2019-05-31 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Mediastinal Lymphoma; Hodgkin Lymphoma; Non Hodgkin Lymphoma
Keywords: Lymphoma; Radiotherapy; Mediastinum; Adverse effects; Longitudinal; Cardiac toxicities; Lung; Breast
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The patients with mediastinal malignant lymphoma: Patients whose radiation therapy field essentially encompasses anterior mediastinum; namely, the majority of malignant lymphoma patients with mediastinal involvement.
  Interventions: Radiation: Standard treatment protocol with combined chemoradiation

INTERVENTIONS:
Radiation: Standard treatment protocol with combined chemoradiation — As for consolidative RT used in patients with early-stage Hodgkin lymphoma, the RT field must essentially include the mediastinum.

SUMMARY:
Malignant anterior mediastinal tumors essentially include lymphomas and thymomas. The location of mediastinum is anatomically close to several critical organs such as heart, lung, and breasts, which might be affected meaningfully when the mediastinal region is irradiated. There have been quite a few studies investigating long-term toxicities concerning the above critical organs and risks of secondary malignancies related to treatment regimens combining chemotherapy and mediastinal radiotherapy. With the advancement of modern radiotherapy, highly conformal and intensity modulated radiotherapy have become a radiotherapeutic standard in recent years. However, most previous studies analyzed patients treated in the era of 2D techniques rather than conformal 3D plans. Almost inevitably, a large volume of the heart and lung was irradiated via the 2D technique with which substantial dose levels might be given to these organs unavoidably. Certainly long-term radiotherapy related toxicities are significantly associated with the dose and volume irradiating the normal organs at risk. Relying on the techniques of modern conformal radiotherapy and the contemporary strategy of multimodality therapy, the dose and volume irradiating the heart and lung were considerably reduced. Therefore, objective tools including heart echocardiography and lung function test will be utilized in this prospective study to evaluate and monitor mainly the patients diagnosed as malignant lymphoma who are recommended to receive mediastinal radiotherapy in the era of modern treatment strategy and techniques.

The participants potentially included in the current study are mainly lymphoma patients with mediastinal malignant lymphoma or patients whose radiation therapy field essentially encompasses anterior mediastinum. Patients are prospectively enrolled in this study after physicians' clinical judgement. After signing the consent form, the recruited patient will receive comprehensive pre-radiotherapy evaluations, including cardiac echocardiography, laboratory tests (BNP, and NT-pro BNP), and lung function tests. Participants who are particularly female patients under the age of 45 will receive pre-radiotherapy breast echocardiography. Radiotherapy treatment planning of both photon and proton respectively will be simulated on Eclipse® treatment planning system. Subsequently participants will receive mediastinal RT within one month after being enrolled in the study. Eligible patients should receive standard multidisciplinary treatment as the tumor board at our institute has suggested. Modern radiotherapy techniques comprise all available modalities in our hospital, including photon or proton beams, intensity-modulated radiotherapy, volumetric modulated arc therapy, image-guidance, and breathing control system. The prescription of treatment field designing and dose scheme will comply with our institutional protocols and updated cancer treatment guidelines. Participants will receive longitudinal follow-up examinations at 3, 6, 9, 12, 18, 24, 36 months after the start of RT course. Standardized examinations include the above mentioned cardiac echocardiography and relevant tests.

It is anticipated that long-term mediastinal RT-related late effects are prospectively and longitudinally surveyed through consistent heart examinations and lung function tests. Long-term effects are expected to be lower with using maturely and widely adopted modern RT techniques. Therapeutic and survival outcomes are expected to be satisfactory, achieving the international level in this prospective observational study focusing on mainly lymphoma patients with mediastinal involvement who are suggested and scheduled to receive mediastinal RT as part of the combined modality treatment.

This study aims to standardize the application of clinical examinations including cardiac echocardiography, lung function tests, and relevant laboratory tests as part of objective tools for monitoring patients' cardiac and pulmonary functions after receiving mediastinal RT. Therefore, it is expected that the risk factors of predisposing patients to develop cardiac toxicities after chemoradiation particularly including mediastinal RT will be explored and identified. In addition objectivity of BNP (or NT-pro BNP) will also be verified in combination with the objective measurement and findings obtained from cardiac echocardiography. It is anticipated that our study would be an important and leading one that integrates radiation oncology, hematology, cardiology, and pulmonology into prospective and longitudinal cardiopulmonary surveillance carried out for mainly malignant lymphoma patients undergoing mediastinal RT in this era of modern chemoradiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an age of more than 15 years old when encountering local radiotherapy
* Histologically confirmed Hodgkin lymphoma or non-Hodgkin lymphoma
* A patient with resected thymoma referred for undergoing postoperative adjuvant radiotherapy is also acceptable and might be feasible
* The intended radiation field should involve the mediastinum region
* Malignant lymphoma patients who have undergone systemic chemotherapy with appropriate intensity and cycles tailored to the histologic subtype and oncological staging should start receiving RT within one month after restaging oncological surveys are performed before the course of mediastinal RT. Patient who must complete standard chemotherapy appropriate for the histologic subtype and staging of lymphoma and also be able to start radiation therapy within one month after restaging oncological surveys performed after completing chemotherapy
* Patients should have a fair to good performance status better than Eastern Cooperative Group (ECOG) of 2.
* Life expectancy of at least 12 months

Exclusion Criteria:

* Pregnant or breastfeeding
* Prior therapeutic radiation therapy delivered to breast, thoracic, or head & neck
* Patients who have a serious medical illness

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The lymphoma patients with mediastinal malignant lymphoma or patients whose radiation therapy field essentially encompasses anterior mediastinum.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in heart function. | 12 month, and 24 month.
  The outcome assessed by cardiac echocardiography. Our study use the standard imaging modality -cardiac echocardiography

SECONDARY OUTCOMES:
Change in cardiac biomarkers. | 1 year, 2 years, 3 years
  The outcome assessed by plasma concentrations of BNP and NT-proBNP
Change in lung function. | 1 year, 2 years, 3 years
  The outcome assessed by lung function test. The lung function tests contain following four tests: "Determination of F. R. C" & "Diffusion capacity rate" & "Screening sporometry before & after B. D." and "Simple bronchodilator test".
Change in cardiac systolic and diastolic functions including left ventricular global longitudinal strain. | 1 year, 2 years, 3 years
  The outcomes assessed by echocardiography
Significant toxicities. | 1 year, 2 years, 3 years
  The outcome assessed by CTCAE v5.0
Disease failure rate within radiation fields | 3 years
Event-free survival | 3 years
Overall survival | 3 years
  Overall survival time, indicated by the time from the date of recruitment to the date of expiring
Progression-Free Survival | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No